CLINICAL TRIAL: NCT01883076
Title: Phase I Safety Study of Autologous Umbilical Cord Blood Derived Mononuclear Cells During Surgical Stage II Palliation of Hypoplastic Left Heart Syndrome
Brief Title: Safety Study of Autologous Umbilical Cord Blood Cells for Treatment of Hypoplastic Left Heart Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy J Nelson, MD, PhD (Other)
Collaborators: University of Oklahoma (Other); Children's Hospital of Philadelphia (Other); Children's Hospitals and Clinics of Minnesota (Other); Children's Hospital Los Angeles (Other); Children's Hospital Colorado (Other); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Timothy J Nelson, MD, PhD, Program Director, ReGen Theranostics, Inc.
Organization: ReGen Theranostics, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-008521
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; HLHS; Congenital Heart Disease; Umbilical cord blood; UCB; Cord blood; Stem cells; Regenerative therapy; Stage II Glenn; Glenn Surgery
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous cell-based delivery (Experimental): autologous cell-based delivery a target dose of 3 million cells / kg of body weight will be delivered into the right heart muscle at the time of surgery. Cells are derived from autologous (self) umbilical cord blood.
  Interventions: Biological: autologous cell-based delivery

INTERVENTIONS:
Biological: autologous cell-based delivery — autologous cells (derived from "self")
  Other Names: umbilical cord blood derived mononuclear cells

SUMMARY:
This is a Phase I study to determine the safety and feasibility of injections of autologous umbilical cord blood (UCB) cells into the right ventricle of Hypoplastic Left Heart Syndrome (HLHS) children undergoing a scheduled Glenn surgical procedure.

The investigators are doing this research study to find out if autologous stem cells from the individual's own umbilical cord blood can be used to strengthen the muscle of the right side of their heart. This will help determine the safety and feasibility of using cell-based regenerative therapy as an additional treatment for the management of HLHS.

DETAILED DESCRIPTION:
This study is a Phase I trial to determine the safety of autologous mononuclear cells (MNC) derived from umbilical cord blood for intramyocardial delivery into the right ventricle during a planned and non-emergent Stage II surgical palliation in subjects with HLHS. This is the first critical step towards applying autologous MNC therapy as an add-on regenerative intervention for congenital heart disease management. The choice of HLHS as the target disease for regenerative therapies in congenital heart disease management is multi-factorial and includes the following considerations: 1) Severity of of this incurable disease, 2) palliative nature and burden of long-term outcomes with a single right ventricular system, 3) three stages of planned surgical procedures that provide time points to adjunctively intervene, and 4) prenatal diagnosis enabling planned collection of UCB. An emerging goal for cardiac regeneration includes the application of cell-based technology to congenital heart disease, which is a favorable substrate due to the lack of fibrotic scaring, and the presence of a microenvironment that is expected to support ongoing cardiac proliferation and growth for functional remuscularization. This Phase I safety study will determine the feasibility of collection, processing, and delivery of autologous cells as used in adult cardiac regenerative protocols in the setting of HLHS surgical management.

ELIGIBILITY:
Inclusion Criteria

1. Individuals with autologous cord blood product that met all cell release criteria (listed on the certificate of analysis from Mayo Clinic Human Cell Therapy Lab) as follows:

   1. No aerobic or anaerobic bacterial growth after 14 days
   2. Greater than 70% cell viability pre-freeze
   3. Total Nucleated Cells (TNC) concentration of 30-42 x 106 cells/mL (pre-freeze)
   4. Minimum of one (1) vial of cells
   5. Mononuclear cell percentage of greater than 50%
   6. Endotoxin result of less than 16 Endotoxin Units (EU)/mL.
2. Mother's serology test results are negative for HIV, Hepatitis B, and Hepatitis C.
3. Individuals with HLHS having undergone Stage I surgical palliation and undergoing planned Stage II palliative Glenn surgery.
4. Ages up to 18 months are eligible if written informed consent can be obtained from both parents (unless one parent is not reasonably available) and/or legal guardians.

Exclusion Criteria

1. Child who's UCB does not meet the specified cell release criteria in Inclusion Criterion #1.
2. History of dimethyl sulfoxide (DMSO) reaction for either the child or mother.
3. Parent(s)/child unwilling to participate.
4. Child with severe chronic diseases, extensive extra-cardiac syndromic features, or history of cancer.
5. Child not completing all pre-procedure work-up within 10 days of the Stage II Glenn surgery as listed in section 6 of this protocol AND lack of pre-procedure work-up documented as a safety concern by a site investigator.
6. Child who's cells have been compromised after meeting cell release criteria (as defined in Inclusion Criterion #1).
7. Child with the following complications of their congenital heart disease:

   1. Any condition requiring urgent, or unplanned procedure within 15 days prior to Stage II surgical repair
   2. Severe pulmonary hypertension (reported in the medical record as >70% systemic pressure)
   3. Other clinical concerns as documented by a site investigator that would predict (more likely to happen than not to happen) a risk of severe complications or very poor outcome during or after Stage II surgical repair.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-05-15 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence of all-cause mortality | Within 2 years following cell therapy treatment
Incidence of new and worsening adverse cardiac events | Within 2 years following cell therapy treatment
  The adverse cardiac events would include sustained/symptomatic ventricular arrhythmias, heart failure, myocardial infarction, cardiac infections, and unexpected cardiovascular surgery.
Percentage of subjects whose cells meet all cell release criteria | Up to 2 years
Percentage of subjects enrolled who undergo cell therapy treatment | Up to 2 years

SECONDARY OUTCOMES:
Change in right ventricular ejection fraction at one month according to cardiac imaging with echocardiography | baseline, 1 month
Change in right ventricular ejection fraction at 3 months according to cardiac imaging with echocardiography | baseline, 3 months
Change in right ventricular ejection fraction at 6 months according to cardiac imaging with echocardiography | baseline, 6 months
Change in right ventricle tricuspid annular plane systolic excursion (TAPSE) at one month according to cardiac imaging with echocardiography | baseline, 1 month
Change in right ventricle TAPSE at 3 months according to cardiac imaging with echocardiography | baseline, 3 months
Change in right ventricle TAPSE at 6 months according to cardiac imaging with echocardiography | baseline, 6 months
Change in right ventricle fractional area change at one month according to cardiac imaging with echocardiography | baseline, 1 month
Change in right ventricle fractional area change at 3 months according to cardiac imaging with echocardiography | baseline, 3 months
Change in right ventricle fractional area change at 6 months according to cardiac imaging with echocardiography | baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Nelson, M.D., Ph.D., Study Director — Mayo Clinic; Muhammad Y Qureshi, MBBS, Principal Investigator — Mayo Clinic; Harold M Burkhart, M.D., Principal Investigator — Oklahoma University Children's Hospital; Joseph W Rossano, M.D., Principal Investigator — Children's Hospital of Philadelphia; David M Overman, M.D., Principal Investigator — Children's Hospital of Minnesota; Ram Kumar Subramanyan, M.D., Ph.D., Principal Investigator — Children's Hospital Los Angeles; James Jaggers, M.D., Principal Investigator — Children's Hospital Colorado
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Oklahoma University Children's Hospital, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials